CLINICAL TRIAL: NCT05111600
Title: Multicentre, Open-label, Uncontrolled, Pivotal Clinical Trial to Confirm the Efficacy and Safety of Autologous Fibrin-cultured Epidermal Grafts Containing Epidermal Stem Cells Genetically Modified for Restoration of Epidermis in Patients With Junctional Epidermolysis Bullosa
Brief Title: Open-label, Pivotal Clinical Trial to Confirm Efficacy and Safety of Autologous Grafts Containing Stem Cells Genetically Modified for Epidermis Restoration in Patients With Junctional Epidermolysis Bullosa
Acronym: HOLOGENE 5
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Development program review and update due to Sponsor re-organization
Sponsor: Holostem s.r.l. (Industry)
Collaborators: IRCCS San Raffaele (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTA-HG5-02
Record Dates: First submitted 2021-09-01; First posted 2021-11-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Junctional Epidermolysis Bullosa Non-Herlitz Type
MeSH Terms: conditions — Epidermolysis Bullosa, Junctional, Non-Herlitz Type | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): After confirmation of eligibility criteria and ICF signature, subject undergoes to skin biopsy for collection of autologous epidermal cells to be used to produce IMP under GMP process. Approximately 2 months later, IMP is transplanted on selected area.
  Interventions: Drug: Transplantation

INTERVENTIONS:
Drug: Transplantation — Implantation of autologous cultured grafts containing genetically modified stem cells for restoration of functional skin on pre-selected areas
  Other Names: Engraftment

SUMMARY:
Prospective, multicenter and multinational, open-label, uncontrolled clinical study to assess the safety and efficacy of autologous cultured epidermal grafts containing epidermal stem cells genetically modified transduced with a LAMB3-gamma retroviral vector. The purpose of this study is to demonstrate the safety and efficacy after one or more treatments with genetically corrected cultured epidermal autograft (Hologene 5) for restoration of the epidermis in patients with generalized intermediate LAMB3-dependent Junctional Epidermolysis Bullosa.

DETAILED DESCRIPTION:
This trial aims to prove the efficacy and safety of RV-LAMB3-transduced epidermal stem cells and lead to a permanent therapy for the skin lesions affecting JEB patients.

Patients are screened according to the Study Inclusion and Exclusion criteria and if found eligible, participants are candidate for the treatment. After confirmation of eligibility, patients will undergo to biopsy for the collection of the autologous epidermal cells used to produce the tissue for the treatment. If all criteria are met, the transplantation of the new cultured transgenic epidermis will be planned according to the procedures and the need of the patient. The study treatment consists of a surgical intervention for new restored stem cells implantation. The surgery is carried out in 2 stages, the first aims at taking biopsy to isolate epidermal cells including stem cells. The biopsy is processed in a laboratory of a regenerative medicine manufacturing site where the tissue is corrected, expanded and prepared as final sheets to be implanted. Afterward, the patient undergoes to the second intervention when the grafts containing genetically corrected cultured keratinocytes (Hologene-5) are implanted into the selected area under local or general anaesthesia.

The treated area is then immobilized for some days after this surgery. Antibiotics and anti-inflammatory drugs may be administered (if necessary) to prevent infections and to minimise swelling.

The follow-up after implantation is 12 months. The treatment can be repeated. The end of the trial is defined as the last visit of the last patient after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-related procedures.
2. Male and female patients between 6 months and 65 years old;
3. Diagnosis of generalized intermediate LAMB3-dependent JEB, confirmed by NGS or Sanger sequencing and/or immunofluorescence;
4. Detectable residual expression of laminin 332 (and its beta-3 chain) by immunofluorescence and/or Western Blot analysis;
5. Presence of blisters and/or ≥ 6 cm2 erosions (persistent or recurrent for more than 3 months); the area of the erosion can be considered as the sum of smaller areas in the same body part (i.e. leg, thigh, arm, …)
6. A cooperative attitude to follow the study procedures (caregivers in case of children);
7. Patients' compliance with the study schedule and procedures, including complete immobilization of the transplanted areas for at least two weeks and hospitalization up to 1 month after transplantation.

Exclusion Criteria:

1. Known or suspected intolerance to anaesthesia;
2. Bad general condition (ECOG index >1);
3. Presence of any skin cancers in the area(s) qualified for treatment;
4. Clinical and/or laboratory signs of acute systemic infections at the time of screening. Patient can be re-screened after appropriate treatment;
5. Female subjects: Pregnant (as evident by a positive urine hCG or serum-hCG test) or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential [WOCBP]) UNLESS they are willing to use highly effective birth control methods;
6. Allergy, sensitivity or intolerance to study medication excipients or other material required by study protocol (as per Investigator's brochure)
7. Contraindications to the local or systemic antibiotics and/or corticosteroids foreseen by the protocol;
8. Contraindications to undergo extensive surgical procedures;
9. Presence of i) systemic diseases, ii) clinically significant or unstable concurrent disease, iii) other concomitant medical conditions, iv) other clinical contraindications to stem cell transplantation, which based on Investigator's judgment, in consultation with the Sponsor Medical Expert may affect the participation in the study or the grafting procedure;
10. Patients (or parents in case of paediatric subject) unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments.
11. Previous treatments or clinical trials envisaging the use of cells (including bone marrow transplantation, BMT) and/or both in vivo or ex vivo gene therapy products.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Re-epithelialization | 12 months
  Re-epithelialization in absence of blisters in at least 50% of the transplanted area measured by the Investigator
Protein residual expression | 12 months
  Protein residual expression resulting in 'Yes' or 'Partial' measured by Immunofluorescence
Expression of transgenic mRNA | 12 months
  Expression of transgenic mRNA resulting in 'Yes' or 'Partial' measured by In situ hybridization
Hemidesmosomes presence | 12 months
  Presence of hemidesmosomes measured by electron microscopy
Skin stability | 12 months
  Negativity or positivity at the stripping test
Patient Reported Outcome | 12 months
  Chnage in Patient Reported Outcome score measured by 5-points Likert scale, where: 1=Definitely Worsened, 2=Slightly Worsened, 3=Unchanged, 4=Slightly Improved, 5=Definitely Improved

SECONDARY OUTCOMES:
Re-epithelialization by Independent Assessor | 12 months
  % of re-epithelialization assessed by the Independent Assessor
Quality of Life improvement | 12 months
  Change in EBDASI (Epidermolysis Bullosa Disease Activity and Scarring Index) skin section score, where Best score=0 and Worse score=120 for Activity and Best score=0 and Worse score=84 for Damage
Treatment-emergent adverse events | 12 months
  Number and % of treatment-emergent adverse events
Serious adverse events | 12 months
  Number and % of serious adverse events
Adverse events of special interest | 12 months
  Number and % of adverse events of special interest
Adverse drug reactions | 12 months
  Number and % of adverse drug reactions

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Magnoni, MD, Surgeon, Principal Investigator — Struttura Complessa di Dermatologia Azienda Ospedaliero Universitaria Policlinico di Modena
Locations (2):
- Hopital Necker-Enfants Malades, Paris, France
- Struttura Complessa di Dermatologia Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

REFERENCES:
- See also: Hologene 5: A Phase II/III Clinical Trial of Combined Cell and Gene Therapy of Junctional Epidermolysis Bullosa — http://links.email.frontiersin.org/ls/click?upn=Dpg5ochww630xh6EMvshS4k2vZe-2Fd8MH-2FVpzt1-2FUQD91C-2FNL5bIclwWnNjv5HD9izZCaOx2V3EtqIs0Ckedw-2F1A-2BcH3PXDfrM3tKsGvB5mOBFA4D4IQsXZBBoywIR8CqP788TC4QjwkjLexp8GkbdobTlDoKSXKIZ4hzFDGy-2BSoPWinVxRUD26SZk4zWlZmIujIlA-2FcuhGtrzCic2TjA6R9WgboLuof6h4bANVfct1-2BR0PaKBaVQpkvKuBSjOwJY97llGsKrkBbQeTFucCWc6XjFbhLpgcO4VwoW0SZPxFOMb0wxr9TxMiyhhXdL-2Fj3ryc_c_Uho53-2BBXHz3IQwFuqmgP8k0vc6XETh9Rxa541lPSMSnGAcDSIwNa63R8LWkU68mnnscH3GsPwiS7GYOTbVFnuLvR-2F6xG6nfgMBA6u57DAAcghHjoQgF1ekrer-2BMmuEgMoSQJ-2Br7xcgVDOTCTOisKEFWCQ14VP684FGXCk8kzV87l0diRwtDJAzg4RRyX46iK-2F7fkoeyDaTJnM3mYt5-2BqgmH9nN2J575hO0RVIJvYWZCkku-2Fsh7f63TYQ3gN2rLlX